CLINICAL TRIAL: NCT02500485
Title: Drug Interaction Study of Henagliflozin and Retagliptin in Healthy Subjects
Brief Title: The Drug-drug Interaction of SHR3824 and SP2086
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR3824-106
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes
Keywords: SHR3824 SP2086 drug-drug interaction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — henagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SHR3824 20mg/SP2086 100mg (Experimental): One 100-mg tablet of SP2086 once daily on Day 1,2,3,4 followed by two 10-mg tablets of SHR3824 once daily on Day 11,12,13,14, followed by one 100-mg tablet of SP2086 and two 10-mg tablets of SHR3824 on Day 15,16,17,18.
  Interventions: Drug: SHR3824, SP2086

INTERVENTIONS:
Drug: SHR3824, SP2086 — One 100-mg tablet of SP2086 once daily on Day 1,2,3,4 followed by two 10-mg tablets of SHR3824 once daily on Day 11,12,13,14, followed by one 100-mg tablet of SP2086 and two 10-mg tablets of SHR3824 on Day 15,16,17,18.
  Other Names: Henagliflozin, Retagliptin

SUMMARY:
The purpose of the study is to investigate the potential interaction between multiple oral doses of SHR3824 and multiple oral doses of SP2086 in healthy adult volunteers.

DETAILED DESCRIPTION:
This is an open-label (volunteers will know the names of treatments they are assigned) single-center study of SHR3824 and SP2086 in healthy adult volunteers. SHR3824(a Sodium-Glucose Cotransporter 2 inhibitor) is currently under development to lower blood sugar levels in patients with type 2 diabetes mellitus (T2DM) ,and SP2086(a Dipeptidyl peptidase IV inhibitor) is also currently under development to lower blood sugar levels in patients with type 2 diabetes mellitus (T2DM).SP2086 will be administered orally (by mouth) as 100mg on Days 1, 2, 3, 4, 15, 16, 17 and 18, SHR3824 will be administered orally (by mouth) as 20mg on Days 11, 12, 13, 14, 15, 16, 17 and 18. Both SHR3824 and SP2086 tablets will be taken with 8 ounces (240 mL) of water.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index (BMI, a measure of a person's weight in relation to height) between 19 and 24 kg/m2.

Exclusion Criteria:

* History of diabetes
* History of heart failure or renal insufficiency,Urinary tract infections, or vulvovaginal mycotic infections
* History of or current clinically significant medical illness as determined by the Investigator
* History of clinically significant allergies, especially known hypersensitivity or intolerance to lactose
* Known allergy to SHR3824 or SP2086 or any of the excipients of the formulation of SHR3824 or SP2086

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of SHR3824. | At protocol-specified times up to Day 14 and Day 18.
  Cmax (a measure of the body's exposure to SHR3824) will be compared before and after administration of multiple doses of SP2086.
The area under the plasma concentration-time curve (AUC) of SHR3824. | At protocol-specified times up to Day 14 and Day 18.
  AUC (a measure of the body's exposure to SHR3824) will be compared before and after administration of multiple doses of SP2086.
The maximum plasma concentration (Cmax) of SP2086. | At protocol-specified times up to Day 4 and Day 18.
  Cmax (a measure of the body's exposure to SP2086) will be compared. before and after administration of multiple doses of SHR3824
The area under the plasma concentration-time curve (AUC) of SP2086. | At protocol-specified times up to Day 4 and Day 18.
  AUC (a measure of the body's exposure to SP2086) will be compared before and after administration of multiple doses of SHR3824.
The number of volunteers with adverse events as a measure of safety and tolerability. | Up tp day 18.

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I Unit of Tongji Hospital affilated Tongji Medical School of Huangzhong Science and Thechnology, Wuhan, Hubei, China